CLINICAL TRIAL: NCT01745211
Title: 755nm Alex Laser for Treatment of Stretch Marks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYN12-PICO-STRIAE_RG4
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Results first posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Striae
MeSH Terms: conditions — Striae Distensae | interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 755nm Alexandrite laser with array handpiece (Experimental): Device: 755nm Alexandrite laser with array handpiece
  Interventions: Device: 755nm Alexandrite Laser

INTERVENTIONS:
Device: 755nm Alexandrite Laser — 755nm Alexandrite laser with array handpiece

SUMMARY:
Evaluate the safety and efficacy of the bilateral treatment of striae using a 755nm Alexandrite laser.

ELIGIBILITY:
Inclusion Criteria

1. Is a healthy male or female between 18 and 85 years old.
2. Has unwanted striae and wishes to undergo laser treatments to remove or improve them.
3. Is willing to consent to participate in the study.
4. Is willing to comply with all requirements of the study including being photographed, following post treatment care and attending all treatment and follow up visits.

Exclusion Criteria

1. Is hypersensitive to light exposure.
2. Has active localized or systemic infection.
3. Is taking medication(s) for which sunlight is a contraindication.
4. Has a history of squamous cell carcinoma or melanoma.
5. Has a history of keloid scarring.
6. Has used oral isotretinoin (Accutane®) within 12 months of initial treatment or plans on using during the course of the study. Note: Skin must regain its normal degree of moisture prior to treatment.
7. Has a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications.
8. Is female and pregnant, has been pregnant within the last 3 months, is currently breast feeding or planning a pregnancy during the study period.
9. Is allergic to lidocaine, tetracaine or Xylocaine with epinephrine.
10. Has any other reason determined by the physician to be ineligible to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- Laser & Skin Surgery Center of New York, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each patient's striation area was treated with the array handpiece. No patients were treated with the standard handpiece.
Units Other Than Participants: striae area
Period: Overall Study
Arm/Group | 755nm Alexandrite Laser
Started | 45; 104 striae area
Completed | 27; 64 striae area
Not Completed | 18; 40 striae area

BASELINE CHARACTERISTICS:
Groups:
- 755nm Alexandrite Laser: 755nm Alexandrite laser (standard handpiece)
  755nm Alexandrite Laser: 755nm Alexandrite laser with modified and standard handpiece
Arm/Group | 755nm Alexandrite Laser
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: African American | 6
  Race/Ethnicity: Asian | 5
  Race/Ethnicity: Hispanic | 9
  Race/Ethnicity: W. Indian | 1
  Race/Ethnicity: Caucasian | 24
Fitzpatrick Skin Score [Count of Participants; unit: Participants] — The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is.
  The scale comes from this source:
  Gupta, Sharma. Skin typing: Fitzpatrick grading and others. Clinics in Dermatology. 2019;37(5):430-436. doi:10.1016/j.clindermatol.2019.07.010
  Participants
    Fitzpatrick Skin Score I | 4
    Fitzpatrick Skin Score II | 9
    Fitzpatrick Skin Score III | 17
    Fitzpatrick Skin Score IV | 9
    Fitzpatrick Skin Score V | 2
    Fitzpatrick Skin Score VI | 4

OUTCOME MEASURES:

1. Primary Outcome: Photographic Evaluation of Striae Clearance
Description: The physician will judge the overall improvement by selecting from improvement ranges of 0-25%, 25-50%, 50-75%, or 75-100% clearance when compared to the baseline.
Time Frame: Follow Up Between 1 and 3 Months Post Last Treatment
Population: 5 subject withdrew and 13 were lost to follow up.
Measure: Count of Units; unit: areas with striation
Units Other Than Participants: areas with striation
Arm/Group | 755nm Alexandrite Laser With Array Handpiece
Number analyzed (Participants) | 27
Number analyzed (areas with striation) | 64
areas with striation
  0-25% Improvement from Baseline | 36
  25-50% Improvement from Baseline | 17
  50-75% Improvement from Baseline | 11

ADVERSE EVENTS:
Time Frame: Adverse events, whether serious or non-serious, were followed throughout study completion, about 18 months.
Groups:
- 755nm Alexandrite Laser: 755nm Alexandrite laser 755nm Alexandrite Laser: 755nm Alexandrite laser with array handpiece
Arm/Group | 755nm Alexandrite Laser
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 26/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 755nm Alexandrite Laser (N=45)
Redness (Skin and subcutaneous tissue disorders) | 23
Crusting (Skin and subcutaneous tissue disorders) | 1
Blistering (Skin and subcutaneous tissue disorders) | 1
Burn (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.